CLINICAL TRIAL: NCT02294539
Title: Comparison of Effects Between Calcium Channel Blocker and Diuretics in Combination With Angiotensin II Receptor Blocker on 24-hr Central Blood Pressure and Vascular Hemodynamic Parameters in Hypertensive Patients Multicenter, Double-blind, Active-controlled, Phase 4 Randomized Trial
Brief Title: Comparison of Effects Between Amlodipine and Hydrochlorothiazide in Combination With Losartan on 24-hr Central Blood Pressure in Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chong-Jin Kim (Other)
Collaborators: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor-Investigator, Chong-Jin Kim, Chairman of Cardiovascular Center, Kyung Hee University Hospital at Gangdong
Organization: Kyung Hee University Hospital at Gangdong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KSH_AMST
Record Dates: First submitted 2014-11-12; First posted 2014-11-19 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Losartan; Amlodipine; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Losartan 50mg/amlodipine 5mg (Experimental): Once daily, 1T, PO medication
  Interventions: Drug: Losartan 50mg/Hydrochlorothiazide 12.5mg
- Losartan 100mg/amlodipine 5mg (Experimental): Once daily, 1T, PO medication
  Interventions: Drug: Losartan 100mg/Hydrochlorothiazide 25mg
- Losartan50 mg/Hydrochlorothiazide12.5 mg (Active Comparator): Once daily, 1T, PO medication
  Interventions: Drug: Losartan 50mg/amlodipine 5mg
- Losartan100 mg/Hydrochlorothiazide25 mg (Active Comparator): Once daily, 1T, PO medication
  Interventions: Drug: Losartan 100mg/amlodipine 5mg

INTERVENTIONS:
Drug: Losartan 50mg/amlodipine 5mg — once daily, 1T, PO medication
  Other Names: amosartan 5/50mg
  Arms: Losartan50 mg/Hydrochlorothiazide12.5 mg
Drug: Losartan 100mg/amlodipine 5mg — once daily, 1T, PO medication
  Other Names: amosartan 5/100mg
  Arms: Losartan100 mg/Hydrochlorothiazide25 mg
Drug: Losartan 50mg/Hydrochlorothiazide 12.5mg — once daily, 1T, PO medication
  Other Names: Cozaar Plus
  Arms: Losartan 50mg/amlodipine 5mg
Drug: Losartan 100mg/Hydrochlorothiazide 25mg — once daily, 1T, PO medication
  Other Names: Cozaar Plus F
  Arms: Losartan 100mg/amlodipine 5mg

SUMMARY:
The purpose of this study is to investigate which combination therapy is more effective for improving the blood pressure (BP) and AM central SBP in hypertensive patients:Angiotensin II receptor blocker (ARB) plus calcium channel blocker (CCB) or ARB plus diuretics

ELIGIBILITY:
Inclusion Criteria:

* Hypertension patients not included exclusion criteria
* Mean seated SBP ≥140mmHg in patients with newly Diagnosed

Exclusion Criteria:

- msDBP≥110mmHg or ms SBP ≥ 180mmHg at the screening and randomization visit

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2014-08; Primary Completion 2016-05-18 (Actual); Study Completion 2016-05-18 (Actual)

PRIMARY OUTCOMES:
change from baseline in msSBP | 4 weeks

SECONDARY OUTCOMES:
change from baseline in AMcSBP | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chong-Jin Kim, Principal Investigator — Kyung Hee University Hospital at Gangdong
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea

REFERENCES:
- [Derived] Cho EJ, Lee HY, Sung KC, Park S, Sohn IS, Park CG, Choi DJ, Ha JW, Ahn YK, Shin J, Hong SJ, Kim SK, Chung WJ, Yoo BS, Hong TJ, Youn HJ, Cho MC, Chae SC, Kim YJ, Kim CJ. Comparison of 24-Hour Ambulatory Central Blood Pressure Reduction Efficacy Between Fixed Amlodipine or Up-Titrated Hydrochlorothiazide Plus Losartan: The K-Central Study. Am J Hypertens. 2019 Sep 24;32(10):992-1002. doi: 10.1093/ajh/hpz050. PMID 31099387
- [Derived] Oh GC, Lee HY, Chung WJ, Youn HJ, Cho EJ, Sung KC, Chae SC, Yoo BS, Park CG, Hong SJ, Kim YK, Hong TJ, Choi DJ, Hyun MS, Ha JW, Kim YJ, Ahn Y, Cho MC, Kim SG, Shin J, Park S, Sohn IS, Kim CJ. Comparison of effects between calcium channel blocker and diuretics in combination with angiotensin II receptor blocker on 24-h central blood pressure and vascular hemodynamic parameters in hypertensive patients: study design for a multicenter, double-blinded, active-controlled, phase 4, randomized trial. Clin Hypertens. 2017 Sep 4;23:18. doi: 10.1186/s40885-017-0074-0. eCollection 2017. PMID 28879040